CLINICAL TRIAL: NCT04803084
Title: Multiparametric MRI as a Non-Invasive Biomarker of the Tumor Microenviroment in Breast Cancer
Brief Title: Multiparametric MRI as a Non-Invasive Biomarker of the Tumor Microenviroment
Status: Suspended | Type: Observational
Why Stopped: MRI upgrade
Sponsor: Laura Kennedy (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Laura Kennedy, Sponsor Investigator, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Other Study IDs: VICC BRE 20104; P50CA098131 (NIH)
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced Pathology: Breast magnetic resonance imaging (MRI) as a preliminary predictive biomarker for breast cancer treatment response.
  Interventions: Other: Tempus assay; Other: Advanced pathology 1; Other: Advanced pathology 2

INTERVENTIONS:
Other: Tempus assay — Blood collection
Other: Advanced pathology 1 — Tissue procurement (from diagnostic biopsy)
Other: Advanced pathology 2 — Tissue procurement (from research biopsy)

SUMMARY:
This study is looking at how an imaging test could help doctors understand if a patient with early breast cancer will respond to drugs that use the patient's immune system to fight cancer.

DETAILED DESCRIPTION:
Primary Objective:

- To evaluate serial multiparametric MRI as an early marker for tumor immune response to an immune checkpoint inhibitor agent

Secondary Objective:

* To assess the potential of early treatment imaging changes on MRI to discern final tumor treatment response
* To assess the prognostic potential of MRI features

Correlative:

* To correlate MRI features with immunophenotypes (i.e. hot and cold tumors)
* To evaluate the association of MRI features with other known biomarkers of immune checkpoint inhibitor response

ELIGIBILITY:
Inclusion Criteria:

Women and men at least 18 years of age.

* Have a new diagnosis of invasive breast cancer with clinical stage I - III disease or regional stage IV with metastasis to the supraclavicular nodes only
* Hormone receptor negative (estrogen-receptor < 5% and/or progesterone-receptor < 5%)
* Human epidermal growth factor receptor 2 (HER2) negative by immunohistochemistry or fluorescence in situ hybridization (FISH)
* Enrollment in a neoadjuvant clinical trial that includes the evaluation of immunotherapy as a part of the regimen; patient must be randomized to a treatment arm (including the control arm) prior to enrolling in this study
* Planning to undergo surgical resection and subsequent adjuvant therapy as per the treatment clinical trial or the clinical provider
* Have tissue available for additional correlative studies OR planned to undergo an additional pre-treatment biopsy for additional tissue acquisition as per provider or the treatment clinical trial
* Be a candidate for MRI imaging.
* Be willing to comply with scheduled visits required for the trial.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Systemic or locoregional treatment for the current episode of breast cancer prior to baseline breast MRI.

* Poor visualization of the tumor on the initial breast MRI (investigator discretion)
* Pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women and men at least 18 years of age that have a new diagnosis of invasive breast cancer with clinical stage I - III disease or regional stage IV with metastasis to the supraclavicular nodes only.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Correlate dynamic-contrast enhanced MRI characteristics | Baseline up to about 14 weeks
Correlate diffusion weight imaging MRI characteristics | Baseline up to about 14 weeks

SECONDARY OUTCOMES:
Evaluate association between MRI features and pathologic response | Baseline up to about 14 weeks
Evaluate association between MRI features and recurrence-free survival | Baseline up to about 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kennedy, MD, PhD, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT04803084/ICF_000.pdf